CLINICAL TRIAL: NCT00113308
Title: A Phase III, 12-Week, Multicentre, Double-Blind, Randomised, Placebo- and Active Comparator-Controlled, Parallel Group Study to Investigate the Efficacy and Safety of GW406381, 5mg, 10mg, 25mg, and 50mg Administered Orally Once Daily, in Adults With Rheumatoid Arthritis
Brief Title: COX-2 Inhibitor Study In Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CXA30009
Record Dates: First submitted 2005-06-07; First posted 2005-06-08 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; COX-2 Inhibitor
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GW406381X

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW406381

SUMMARY:
This study is being conducted to find out if an investigational drug called GW406381 can help people with rheumatoid arthritis.

ELIGIBILITY:
Inclusion criteria:

* Rheumatoid arthritis (RA) for at least 12 months.
* Required a non-steroidal anti-inflammatory drug (NSAID) or COX-2 inhibitor for RA for at least 5 out of 7 days of each week for the 4 weeks prior to screening.

Exclusion criteria:

* Any history of cardiovascular disease (e.g., heart attack, stroke, congestive heart failure, uncontrolled high blood pressure), documented peripheral arterial insufficiency and symptomatic, clinically significant claudication, or who have a history of peripheral arterial embolism.
* Have an active stomach ulcer or history of any stomach tear or bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2208 (Actual)
Dates: Start 2005-06; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Percentage of American College of Rheumatology (ACR)20 Responders at Week 12 | Week 12

SECONDARY OUTCOMES:
Change from baseline to each scheduled visit in tender/painful joint count (68 joint panel) | Baseline and Week 12
Change from baseline to each scheduled visit in swollen joint count (66 joint panel) | Baseline and Week 12
Change from baseline to each scheduled visit in patient's pain assessment (VAS) | Baseline and Week 12
Change from baseline to each scheduled visit in physician's global assessment of arthritis condition | Baseline and Week 12
Change from baseline to each scheduled visit in patient's global assessment of arthritis condition | Baseline and Week 12
Change from baseline to each scheduled visit in functional disability index (HAQ) | Baseline and Week 12
Change between baseline and end of treatment (or early withdrawal) in the Short Form - McGill Pain Questionnaire (SF-MPQ) | Baseline and Up to Week 12
Change from baseline to each scheduled visit in C-reactive protein (CRP) | Baseline and up to Week 12
Number of participants withdrawing from the study due to lack of efficacy | Week 12
Number of participants who received supplementary analgesic therapy | Week 12
Changes from pretreatment to on treatment and post-treatment follow-up in vital signs- systolic blood pressure (SBP) and diastolic blood pressure (DBP) | Baseline and up to Week 12
Changes from pretreatment to on treatment and post-treatment follow-up in vital signs- heart rate (HR) | Baseline and up to Week 12
Changes from pretreatment to on treatment and post-treatment follow-up in weight | Baseline and Week 12
Number of participants with change in BMI of potential clinical concern | Week 4, 4, 8, 12 and foloow up
Number of participants with change from baseline of pedal oedema (including diuretic use) | Baseline and up to Week 12
Change from baseline in 12-lead electrocardiograms (ECGs) | Baseline and up to Week 12
Change from baseline in clinical chemistry parameters: Albumin | Baseline and up to Week 12
Change from baseline in clinical chemistry parameters: Alkaline Phosphatase, Alanine Amino Transferase, Aspartate Amino Transferase | Baseline and Up to Week 12
Change from baseline in clinical chemistry parameters: Total Bilirubin | Baseline and up to Week 12
Change from baseline in clinical chemistry parameters: Carbon Dioxide content /Bicarbonate, Glucose, Potassium, Sodium | Baseline and up to Week 12
Change from baseline in clinical chemistry parameters: Creatinine | Baseline and up to Week 12
Change from baseline in haematology parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, Platelet count, White Blood Cell count | Baseline and up to Week 12
Change from baseline in haematology parameters: Hemoglobin | Baseline and up to Week 12
Change from baseline in haematology parameters: Mean Corpuscle volume | Baseline and Up to Week 12
Change from baseline in haematology parameters: Red Blood Cell count | Baseline and up to Week 12
Urinalysis assessment | Up to Week 12
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Upto Week 12
Change in the Short Form-36 (SF-36v2) subscale scores between baseline and the end of treatment (or early withdrawal) | Baseline and Week 12
Change in the Short Form-36 (SF-36v2) Physical component summary score and mental component summary score between baseline and the end of treatment (or early withdrawal) | Baseline and Week 12
Psychometrically test and validate the amended Patient Satisfaction with Pain Medication questionnaire | Week 12
Change between baseline and end of treatment (or early withdrawal) in the EuroQoL Questionnaire -5 Dimensions (EQ-5D) utility score, using European population utility tariff | Baseline and Week 12
Change between baseline and end of treatment (or early withdrawal) in the fatigue/inertia factor of the Profile of Moods States Brief Form (POMS-B) | Baseline and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (276):
- United States (88):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Montgomery, Alabama
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Palm Desert, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Bridgeport, Connecticut
  - GSK Investigational Site, Danbury, Connecticut
  - GSK Investigational Site, Hamden, Connecticut
  - GSK Investigational Site, Trumbull, Connecticut
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Dunedin, Florida
  - GSK Investigational Site, Largo, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Palm Harbor, Florida
  - GSK Investigational Site, Port Orange, Florida
  - GSK Investigational Site, Stuart, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Trinity, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Zephyrhills, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Gainsville, Georgia
  - GSK Investigational Site, Roswell, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Idaho Falls, Idaho
  - GSK Investigational Site, Evanston, Illinois
  - GSK Investigational Site, Morton Grove, Illinois
  - GSK Investigational Site, Springfield, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Prairie Village, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Slidell, Louisiana
  - GSK Investigational Site, Wheaton, Maryland
  - GSK Investigational Site, Fall River, Massachusetts
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Lansing, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Reno, Nevada
  - GSK Investigational Site, Dover, New Hampshire
  - GSK Investigational Site, Berlin, New Jersey
  - GSK Investigational Site, Mercerville, New Jersey
  - GSK Investigational Site, Johnson City, New York
  - GSK Investigational Site, Kingston, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, North Massapequa, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Gastonia, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Statesville, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Concinnati, Ohio
  - GSK Investigational Site, Mayfield Village, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Duncansville, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, West Reading, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Hampton, South Carolina
  - GSK Investigational Site, Murrells Inlet, South Carolina
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Everett, Washington
  - GSK Investigational Site, Vancouver, Washington
  - GSK Investigational Site, Racine, Wisconsin
- Argentina (7):
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Quilmes
  - GSK Investigational Site, San Juan
  - GSK Investigational Site, San Miguel de Tucumán
- GSK Investigational Site, Vienna, Austria
- Belgium (4):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Diepenbeek
  - GSK Investigational Site, Lommel
  - GSK Investigational Site, Mons
- Bulgaria (3):
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- Canada (14):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Penticton, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Kitchener, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Saint-Jérôme, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
  - GSK Investigational Site, Saskatoon, Saskatchewan
- Chile (2):
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- GSK Investigational Site, San José, Costa Rica
- Denmark (4):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Ishøj
  - GSK Investigational Site, Odense C
  - GSK Investigational Site, Vejle
- Finland (3):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Hyvinkää
  - GSK Investigational Site, Kuopio
- France (9):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Cahors
  - GSK Investigational Site, Chilly-Mazarin
  - GSK Investigational Site, Corbeil-Essonnes
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Tours
- Germany (41):
  - GSK Investigational Site, Baden-Baden, Baden-Wurttemberg
  - GSK Investigational Site, Deggingen, Baden-Wurttemberg
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Kippenheim, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Bayreuth, Bavaria
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Passau, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Hüttenberg, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Einbeck, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Hildesheim, Lower Saxony
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Aachen, North Rhine-Westphalia
  - GSK Investigational Site, Beckum, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Hattingen, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Saarbrücken, Saarland
  - GSK Investigational Site, Chemnitz, Saxony
  - GSK Investigational Site, Delitzsch, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Freital, Saxony
  - GSK Investigational Site, Görlitz, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Schmiedeberg, Saxony
  - GSK Investigational Site, Wolmirstedt, Saxony-Anhalt
  - GSK Investigational Site, Elmshorn, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Pinneberg, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
- Greece (2):
  - GSK Investigational Site, Kavala
  - GSK Investigational Site, Thessaloniki
- Hungary (2):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Győr
- India (6):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Hyderabad, Andhra Pradesh
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Pune
- Ireland (2):
  - GSK Investigational Site, Dublin
  - GSK Investigational Site, Waterford
- Italy (10):
  - GSK Investigational Site, Pescara, Abruzzo
  - GSK Investigational Site, Benevento, Campania
  - GSK Investigational Site, Telese Terme (BN), Campania
  - GSK Investigational Site, Arenzano (GE), Liguria
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Rozzano (MI), Lombardy
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Prato, Tuscany
  - GSK Investigational Site, Terni, Umbria
  - GSK Investigational Site, Montebelluna (TV), Veneto
- Latvia (3):
  - GSK Investigational Site, Liepāja
  - GSK Investigational Site, Riga
  - GSK Investigational Site, Valmiera
- Mexico (4):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, México
- Netherlands (6):
  - GSK Investigational Site, Etten-Leur
  - GSK Investigational Site, Gouda
  - GSK Investigational Site, Heerlen
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Zwolle
- New Zealand (4):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Lower Hutt
  - GSK Investigational Site, Rotorua
- Norway (5):
  - GSK Investigational Site, Harstad
  - GSK Investigational Site, Levanger
  - GSK Investigational Site, Lillehammer
  - GSK Investigational Site, Skien
  - GSK Investigational Site, Tønsberg
- Peru (3):
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, Callao
  - GSK Investigational Site, Lima
- GSK Investigational Site, Manila, Philippines
- Poland (4):
  - GSK Investigational Site, Grudziądz
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- GSK Investigational Site, Caguas, Puerto Rico, Puerto Rico
- Romania (2):
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
- Russia (7):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Tula
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg
- South Africa (10):
  - GSK Investigational Site, Korsten, Eastern Cape
  - GSK Investigational Site, Boksburg, Gauteng
  - GSK Investigational Site, Muckleneuk, Gauteng
  - GSK Investigational Site, Parktown, Gauteng
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Erasmus Kloof, Pretoria
  - GSK Investigational Site, Kempton Park
  - GSK Investigational Site, Observatory
  - GSK Investigational Site, Pinetown
- South Korea (3):
  - GSK Investigational Site, Anyang-si
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Seoul
- Spain (14):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Baracaldo/Vizcaya
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Mérida (Badajoz)
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, San Sebastián
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Villajoyosa
- Ukraine (4):
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lviv
- United Kingdom (6):
  - GSK Investigational Site, Truro, Cornwall
  - GSK Investigational Site, St Albans, Hertfordshire
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, Metropolitan Borough of Wirral, Merseyside
  - GSK Investigational Site, Ashford, Middlesex
  - GSK Investigational Site, Northampton, Northamptonshire